CLINICAL TRIAL: NCT06274905
Title: Topical Anaesthesia in Cutaneous Head and Neck Surgery: a Randomized Controlled Trial
Brief Title: Topical Anaesthesia in Cutaneous Head and Neck Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital Waterford (Other)
Responsible Party: Principal Investigator, Rory O'Neill, Principal Investigator, University Hospital Waterford
Allocation: Randomized | Model: Sequential | Masking: Single | Purpose: Treatment
Other Study IDs: 160123
Record Dates: First submitted 2024-01-27; First posted 2024-02-23 (Actual); Last update posted 2024-02-23 (Actual); Status verified 2024-02

CONDITIONS: Pain, Acute; Head and Neck Cancer; Cutaneous Tumor
MeSH Terms: conditions — Acute Pain; Head and Neck Neoplasms; Skin Neoplasms | interventions — Ethyl Chloride

STUDY DESIGN:
Who Masked: Participant
Masking Description: Single blinding (for participants) only for patients receiving EMLA or EMLA placebo.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- EMLA cream (Experimental): EMLA cream 5% 25g lidocaine, 25g prilocaine; Astra Zeneca. Topically applied followed by Tegaderm dressing to cover. Length of duration monitored and recorded as part of study
  Interventions: Drug: EMLA
- EMLA placebo (Placebo Comparator): Aqueous cream ((Ultrapure Laboratories®️, Mayo, Ireland) applied topically followed by covering with Tegaderm dressing. Length of duration monitored and recorded as part of study
  Interventions: Drug: Aqueous cream BP
- Ethyl chloride spray (Experimental): Ethyl chloride spray (Cryogesic®, Fannin Ltd, Dublin, Ireland). Applied topically to surgical site prior to LA injection. Spray at distance of 5-10cm for 4-8 seconds until skin slightly blanched and the fluid allowed to evaporate.
  Interventions: Drug: Ethyl chloride
- Control group (No Intervention): No intervention administered

INTERVENTIONS:
Drug: EMLA — EMLA cream
  Arms: EMLA cream
Drug: Ethyl chloride — Ethyl chloride
  Arms: Ethyl chloride spray
Drug: Aqueous cream BP — Aqueous cream
  Arms: EMLA placebo

SUMMARY:
This study aims to assess if EMLA or ethyl chloride spray are effective in reducing the pain associated with local anaesthetic administration in cutaneous surgery of the head and neck compared to a placebo and control group through a randomized control trial study design.

DETAILED DESCRIPTION:
Operations on cutaneous tissues of the head and neck are some of the most frequently performed types of operation performed. They can often successfully be performed using local anaesthetic (LA). However, tissues in this anatomic area are some of most sensitive tissues in the body to nociceptive pain. As such, local anaesthetic can be a distressing experience for patients in many ways. Unfortunately, it is also the most common anatomical site for cutaneous malignancies. The majority of these lesions are resected under local anaesthetic. However, one of the major disadvantages of local anaesthetic such as lidocaine is pain during administration.

Several interventions have been used to reduce pain from needles and injections including ethylene chloride cryoanalgesic spray and topical anaesthetic agents including EMLA (lidocaine and prilocaine) and Ametop ointments. These have been extensively used in paediatric populations with great success to reduce pain during procedures requiring hypodermics such as cannulation. Several studies have trialled these interventions in adult populations across a variety of anatomical locations with variable results. The investigators aim to assess the efficacy of EMLA and ethyl chloride in mitigating nociceptive pain associated with local anaesthetic administration in patients undergoing cutaneous head and neck surgery.

ELIGIBILITY:
Inclusion Criteria:

* Aged at least 18 years
* Receiving surgery to cutaneous tissues of the head and neck
* Procedure performed under local anaesthetic

Exclusion Criteria:

* Paediatric patients
* Surgery performed under general anaesthetic
* Mucosal operative site (e.g. oral cavity)
* Significant cognitive impairment (e.g. severe dementia)
* Known sensitivity/allergy to EMLA
* History of a pain disorder (e.g. complex regional pain syndrome).

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 124 (Actual)
Dates: Start 2023-02-20 (Actual); Primary Completion 2023-07-07 (Actual); Study Completion 2023-07-07 (Actual)

PRIMARY OUTCOMES:
Pain score | The pain score is measured essentially immediately after administration of the local anaesthetic (within 20 seconds of administration).
  The primary outcome measure is patient reported pain on a numeric rating scale (NRS)(1; no pain, 10; worst pain imaginable) recorded after LA administration

SECONDARY OUTCOMES:
Patient satisfaction | The overall patient satisfaction score is measured essentially immediately after the operation had concluded (within 20 seconds of completion).
  Patient satisfaction measured on NRS scale of 1=not bad at all, to 10=worst experience imaginable recorded immediately postoperatively

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital Waterford, Waterford, Ireland

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-12-20): https://cdn.clinicaltrials.gov/large-docs/05/NCT06274905/Prot_SAP_000.pdf